CLINICAL TRIAL: NCT04303910
Title: An Analysis of Blood Management in Patients Having Hip or Knee Arthroplasty in Siriraj Hospital: a Retrospective Study
Brief Title: An Analysis of Blood Management in Patients Having Hip or Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Assoc Prof, Siriraj Hospital
Other Study IDs: SIRB421_2
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Transfusion-dependent Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to examine the transfusion rate and appropriateness in patients undergoing elective knee and hip replacement surgery at Siriraj Hospital

DETAILED DESCRIPTION:
The main objective of this study is to examine the transfusion rate and appropriateness in patients undergoing elective knee and hip replacement surgery at Siriraj Hospita by reviewing data from previous medical records (retrospective chart review).

ELIGIBILITY:
Inclusion Criteria:

* Patients Having elective Hip or Knee Arthroplasty in Siriraj Hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients Having elective Hip or Knee Arthroplasty in Siriraj Hospital
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Perioperative transfusion rate | 1 week
  Transfusion rate in Patients Having Hip or Knee Arthroplasty in Siriraj Hospital

SECONDARY OUTCOMES:
Inappropriate transfusion rate | 1 week
  Perioperative inappropriate transfusion rate in Patients Having Hip or Knee Arthroplasty in Siriraj hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No